CLINICAL TRIAL: NCT00392145
Title: Emergency Department Rapid Intravenous Rehydration (RIVR) for Pediatric Gastroenteritis: A Randomized Controlled Trial
Brief Title: Emergency Department Rapid Intravenous Rehydration (RIVR) for Pediatric Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000008579
Record Dates: First submitted 2006-06-27; First posted 2006-10-25 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis; Dehydration
Keywords: Pediatrics; Gastroenteritis; Dehydration; IV Rehydration
MeSH Terms: conditions — Gastroenteritis; Dehydration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Standard IV rehydration
- 2 (Experimental)
  Interventions: Drug: Rapid intravenous rehydration (RIVR)

INTERVENTIONS:
Drug: Standard IV rehydration — A 20 mL/kg 0.9% normal saline bolus (maximum 999 mL) will be administered over 1 hour. This will be followed by D5-0.9% normal saline at a maintenance rate (maximum 55 mL/hr).
  Arms: 1
Drug: Rapid intravenous rehydration (RIVR) — A 60 mL/kg 0.9% normal saline bolus (maximum 999 mL) over 1 hour will be administered. This will be followed by D5-0.9% normal saline at a maintenance rate (maximum 55 mL/hr).
  Arms: 2

SUMMARY:
This study will look at children with dehydration secondary to gastroenteritis requiring IV rehydration and determine whether the proportion rehydrated after two hours is greater in the children who receive rapid intravenous rehydration (RIVR) or in the children who receive standard IV rehydration.

DETAILED DESCRIPTION:
Despite a movement toward increased use of enteral rehydration, many children still receive prolonged IV rehydration in the emergency department (ED). These children commonly receive a single IV bolus of normal saline followed by the administration of a hypotonic solution at a maintenance rate.

The mean time spent in the ED by children receiving IV rehydration is significantly longer than the mean time required to treat all other conditions. ED overcrowding has been associated with poor outcomes, prolonged pain and suffering, and dissatisfaction. One of the solutions proposed in the American Academy of Pediatrics Policy Statement on ED overcrowding is that hospitals should strive to improve the efficiency of the care provided. One small step in this direction may be to improve our management of gastroenteritis and dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Acute gastroenteritis as determined by the supervising physician.
* Age greater than 90 days
* Dehydrated and unable to consume sufficient oral fluids to overcome their dehydration state

Exclusion Criteria:

* Weight less than 5 kg or greater than 33 kg
* Underlying disease which may limit the amount of IV fluids given,including but not limited to: hypoalbuminemic states, renal insufficiency, heart disease requiring pharmacotherapy or lesions that may predispose to congestive heart failure, hypertension, chronic lung disease (excluding asthma), diabetes mellitus, severe anemia, and chronic inflammatory disease
* Clinical suspicion by the attending physician of myocarditis or previously undiagnosed cardiac or renal disease.
* History of abdominal surgery or concern regarding an acute surgical abdomen
* Significant head, chest or abdominal trauma within the preceding 7 days
* Bilious or bloody vomitus
* Evidence of hemodynamic compromise (BP < 80 + 2 * age (yrs)) requiring > 20 mL/kg 0.9% normal saline to be administered in the 1st hour
* Bedside glucose < 2.8 mmol/L (see Section 8.3)
* Unable to provide a telephone number or unavailable for follow-up
* Previously enrolled in this trial

Ages: 90 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2006-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rehydration criteria defined by: dehydration score ≤ 1, normal capillary refill time, normal skin turgor, normal respiratory rate | 2 hours following the initiation of IV rehydration

SECONDARY OUTCOMES:
Hospitalization | 72 hours
Ability to tolerate oral rehydration | Measured per 2 hour time period after consuming 5 mL/kg of liquid
Repeat ED visit | 72 hours
Time (in minutes) from initiation of IV rehydration until disposition determination | Determined by outcome
Attending physician discharge comfort level | Two and four hours following initiation of IV rehydration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Freedman, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Freedman SB, DeGroot JM, Parkin PC. Successful discharge of children with gastroenteritis requiring intravenous rehydration. J Emerg Med. 2014 Jan;46(1):9-20. doi: 10.1016/j.jemermed.2013.04.044. Epub 2013 Aug 30. PMID 23993936
- [Derived] Freedman SB, Parkin PC, Willan AR, Schuh S. Rapid versus standard intravenous rehydration in paediatric gastroenteritis: pragmatic blinded randomised clinical trial. BMJ. 2011 Nov 17;343:d6976. doi: 10.1136/bmj.d6976. PMID 22094316